CLINICAL TRIAL: NCT02017288
Title: Natural History Of Oral Cancer Precursor Lesions: A Prospective Cohort Study
Brief Title: Study to Evaluate the Natural History of Head and Neck Cancer Precursors in Taiwan
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: National Taiwan University (Other); Academia Sinica, Taiwan (Other); China Medical University, China (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999914018; 14-C-N018
Record Dates: First submitted 2013-12-19; First posted 2013-12-20 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Head and Neck Neoplasms
Keywords: Head and Neck Cancers; Larynx; Oropharynx; Oral Cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Laryngeal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- Cancer: Participants diagnosed with incident oral cancer
- Control: Participants without oral lesions or cancers matched to oral cancer/precursor participants on age, gender, smoking/betel nut habits
- Precursor: Participants clinically diagnosed with oral lesions

SUMMARY:
Background:

- Cancer of the mouth and throat is one of the most common cancers in Taiwan. This cancer develops over several years, beginning as white or red patches in the mouth or throat that become growths. It can also cause a condition that leads to rigidity of the cheeks. The growths can be identified when a doctor looks into a person s mouth. It is currently not clear why some people with abnormal growths progress to cancer while others do not. Researchers want to better understand why some patients with early abnormal growths get late abnormal growths. They also want to understand why some people get abnormal growths again, even after they receive treatment.

Objectives:

- To understand why some people with precancerous lesions in their mouth develop cancer while others do not.

Eligibility:

- Adults 21 years and older, some with abnormal growths in the mouth, some without any, and some with head and neck cancer.

Design:

* Participants will visit a hospital in Taiwan 2 times.
* At the first visit, participants will answer questions about their health, lifestyle, and family medical history. A doctor will examine the participant s mouth and take a small piece of any growth they see. They will do this with a brush. They will also photograph the participant s mouth. Participants will also give blood and saliva samples, plus a small sample of a mouth rinse.
* Participants who are diagnosed with a late abnormal growth that is not cancer will return for a second visit. They will answer the same questions and undergo the same procedures as at the first study.

DETAILED DESCRIPTION:
Oral cancers are ideal candidates for screening, early detection, and secondary prevention given the amenability for visual inspection and specimen collection and the availability of recognized precursors. Yet, there are currently no guidelines for screening, treatment, or follow-up of patients with oral cancer precursors, in part, owing to the current gaps in knowledge regarding the natural history of precursor lesions. We propose to conduct a prospective cohort study of patients with oral cancer precursors to address these knowledge gaps and to investigate novel etiologic factors.

In preparation for the cohort study, we recently conducted a pilot study in Taiwan, a country with high oral cancer incidence. This pilot was aimed to streamline field operations and collect preliminary data to aid in the design of the cohort study. As detailed in our concept, we successfully accomplished all of the goals of our pilot study, including successful recruitment and retention of patients as well as the collection of critical preliminary data.

Based on these efforts, we are seeking approval to conduct a prospective cohort study of 3000 patients with precursors to investigate the natural history of histologically-defined oral cancer precursor lesions and evaluate epidemiologic/ molecular predictors for progression. After completion of the recruitment period, we plan to recruit an additional 500 patients with clinically-defined precancerous lesions for passive follow-up. The prospective component will be complemented by cross-sectional comparisons of epidemiologic/molecular factors across 750 controls, 3500 precursors, and 750 cancers.

ELIGIBILITY:
* INCLUSION CRITERIA

We plan to recruit all patients (controls, precursors, and invasive cancers) at the aforementioned two hospitals. Doctors at these hospitals conduct routine visual and tactile examination as part of Taiwan s national oral cancer screening program. For this screening program, all individuals aged 21 years or older who chew betel-quid or smoke are screened through visual inspection for the presence of precursor lesions or cancer.

EXCLUSION CRITERIA

Participants younger than 21 years and individuals with a history of head and neck cancer will be excluded from the study.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A prospective cohort study of 3000 patients with precursors to investigate the natural history of histologically-defined oral cancer precursor lesions and evaluate epidemiologic/ molecular predictors for progression. This prospective component will be complemented by cross-sectional comparisons of epidemiologic/molecular factors across 750 controls, 3000 precursors, and 750 cancers.
Sampling Method: Non-Probability Sample
Enrollment: 3576 (Actual)
Dates: Start 2013-11-18 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
Progression to dysplasia/cancer in participants with oral precursors. | Follow-up visits every 6 months for 5 years
  Histologically confirmed progression to dysplasia/cancer in participants with oral precursors.

CONTACTS AND LOCATIONS:
Overall Officials: Anil K Chaturvedi, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (4):
- Taiwan (4):
  - Chang Gung Memorial Hospital - Kaohsiung, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital- Taoyuan, Taoyuan District